CLINICAL TRIAL: NCT05988216
Title: A Clinical Study on the Safety and Efficacy of BRL-301 (Allogeneic Chimeric Antigen Receptor T Cell Injection Targeting CD19 Gene) in the Treatment of Refractory Systemic Lupus Erythematosus
Brief Title: Universal CAR-T Cells (BRL-301) in Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BRL-301A-SLE-IIT
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRL-301 (Experimental): Allogeneic CD19-targeted Chimeric AntigenReceptor (CAR) T Cells
  Interventions: Biological: BRL-301

INTERVENTIONS:
Biological: BRL-301 — Single dose of Allogeneic Anti-CD19 CAR T cells will be infused
  Other Names: Allogeneic Anti-CD19 CAR T cells

SUMMARY:
This is an investigator initiated trial to assess the efficacy and safety of BRL-301 in the refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
The study had the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 65 years old (including threshold), regardless of gender;
2. Subjects diagnosed with SLE according to the 2019 EULAR/ACR SLE classification criteria; ANA ≥ 1:80, or positive for anti dsDNA and/or anti Sm antibodies;
3. The condition becomes active again after conventional treatment is ineffective or the disease relapses. Conventional treatment is defined as the use of two or more drugs, including corticosteroids (more than 1mg/kg/d) and any one or more of the following immunomodulatory drugs for over six months: antimalarial drugs, cyclophosphamide, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biologics including rituximab, belimumab, etanercept, etc.
4. At least one BILAG2004 Class A or two Class B score, or both;
5. SELENA-SLEDAI score ≥ 8 points;
6. The positive expression and expression rate of CD19 on peripheral blood B cells determined by flow cytometry;
7. The functions of important organs meet the following requirements:

   Bone marrow function needs to meet:
   1. White blood cell count ≥ 3 × 109/L;
   2. Neutrophil count ≥ 1 × 109/L (no Colony-stimulating factor treatment within 2 weeks before examination);
   3. Platelets ≥ 50 × 109/L;d. Hemoglobin ≥ 80g/L

   Liver function:
   1. Alanine Aminotransferase (ALT) ≤ 3 × ULN;
   2. Asparagus cochinchinensis transase (AST) ≤ 3 × ULN;
   3. Total Bilirubin (TBIL) in serum ≤ 1.5 × ULN (excluding Gilbert syndrome, total bilirubin ≤ 3.0 × ULN); Renal function: Creatinine Clearance Rate (CrCl) ≥ 60 ml/minute (Cockcroft/Fault formula) ;

   Coagulation function:
   1. International Normalized Ratio (INR) ≤ 1.5 × ULN,
   2. Prothrombin time (PT) ≤ 1.5 × ULN.

   Cardiac function: good hemodynamic stability, left ventricular Ejection fraction (LVEF) ≥ 55%;
8. Female patients of childbearing potential and male patients whose female sexual partners are of childbearing age should adopt medically recognized contraceptive measures or abstain from sex within at least 6 months after infusion of BRL-301; female patients of childbearing age should have a negative serum HCG test result within 7 days before study enrollment and be not breastfeeding;
9. Willing to participate in this clinical study, sign an ICF, and complete follow-ups, with good compliance.

Exclusion Criteria:

1. Have a serious history of Drug allergy or allergic constitution;
2. Fungi, bacteria, viruses, or other infections that are uncontrollable or require intravenous medication treatment exist or are suspected;
3. Active central nervous system disease caused by SLE or not (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system Vasculitis);
4. Individuals with relatively serious heart diseases, such as angina pectoris, myocardial infarction, heart failure, and arrhythmia;
5. Subjects with congenital immunoglobulin deficiency;
6. Other malignant tumors (excluding non Melanoma skin cancer, cervical cancer in situ, bladder cancer cancer and breast cancer that have survived for more than 5 years without disease);
7. Subjects with end-stage renal failure;
8. Have received any of the following SLE treatments:

   1. Corticosteroid (defined as prednisone or equivalent>20 mg/day) of therapeutic dose were used before enrollment or within 72 hours before BRL-301 infusion.
   2. Use any other clinical study drugs for SLE within 4 weeks prior to enrollment. However, if the research treatment period is ineffective or the disease progresses, and at least 3 half-lives have passed before enrollment, enrollment is allowed.
   3. Had received anti CD20 monoclonal antibody (such as Rituximab) within 4 weeks before screening, tetaximab within 6 weeks, or belizumab within 12 weeks.
   4. Previous CAR-T cell or other genetically modified T Cell therapy.
9. Subjects with positive hepatitis B B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and HBV DNA titer in peripheral blood higher than the upper limit of detection; Patients with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; People who are positive for human immunodeficiency virus (HIV) antibodies; Those who have tested positive for syphilis;
10. Having mental illness and severe cognitive impairment;
11. Those who have participated in other clinical trials within the first 3 months of enrollment;
12. Pregnant or intending to conceive women;
13. Patients who are unsuitable for being included into this study as deemed by the investigator due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The safety of BRL-301 in refractory systemic lupus erythematosus | 3 months
  Incidence and severity of AEs and SAEs, including changes in laboratory values, ECG and vital signs as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
The efficiency of BRL-301 in refractory systemic lupus erythematosus | 3 months
  Number of patients with SRI-4 response: including SELENA-SLEDAI ≥4-Point improvement, BILAG 2004 with No new A domain score AND no more than 1 new B domain scores, PGA with No worsening (<0.3-point increase)
Cellular kinetics | 3 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No